CLINICAL TRIAL: NCT06897527
Title: Phase 4, Open Label, Non-comparative, Interventional, Multicenter Study to Evaluate the Safety of Dostarlimab in Adult Patients in India With Mismatch Repair Deficient (dMMR)/Microsatellite Instability-high (MSI-H) Recurrent or Advanced Endometrial Cancer (EC) That Has Progressed on or Following Prior Treatment With a Platinum-containing Regimen
Brief Title: A Study to Evaluate the Safety of Dostarlimab in Adult Participants in India With Recurrent or Advanced Endometrial Cancer (EC)
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 221460
Record Dates: First submitted 2025-03-20; First posted 2025-03-27 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Neoplasms, Endometrial
Keywords: Dostarlimab; Endometrial cancer; dMMR; MSI-H
MeSH Terms: conditions — Endometrial Neoplasms | interventions — dostarlimab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Dostarlimab (Experimental)
  Interventions: Drug: Dostarlimab

INTERVENTIONS:
Drug: Dostarlimab — Dostarlimab will be administered.

SUMMARY:
The goal of this study is to evaluate the safety profile of dostarlimab in Indian adults with recurrent or advanced endometrial cancer.

ELIGIBILITY:
Inclusion Criteria:

* Participants ≥18 years of age, at the time of signing the informed consent.
* Documented case of dMMR/MSI-H recurrent or advanced EC that has progressed on or following prior treatment with platinum containing regimen.
* Eligible for dostarlimab treatment according to the approved prescribing information and the investigator's clinical judgement.
* WOCBP (Women of childbearing potential) agree to use contraceptive from screening through at least 120 days after the last dose.
* Negative serum or urine pregnancy test at most 72 hours prior to the first dose of study medication.
* Capable of giving signed informed consent which includes compliance with the requirements and restrictions listed in the informed consent form (ICF) and in this protocol, in accordance with applicable laws.

Exclusion Criteria:

* Known active hepatic disease, End-Stage Renal Disease (ESRD) or known case of serious, uncontrolled medical disorder/active infections which precludes participant's inclusion in the study as per the investigator's judgement.
* Either the history of hypersensitivity to excipients of the study drug or to drugs with a similar chemical structure or class of the study drug.
* Received prior therapy with an anti- programmed death receptor 1 (anti-PD-1), anti-PD-1- ligand-1 (anti-PD-L1) agent.
* Has a diagnosis of immunodeficiency or is receiving systemic steroid therapy or any other form of immunosuppressive therapy within 7 days prior to the first dose of study treatment.
* Received a live vaccine within 14 days of planned start of study therapy.
* Participation in another clinical study with a study drug administered in the last 3 months.
* Pregnant, breastfeeding, or expecting to conceive while receiving study treatment and for up to 120 days after the last dose of study treatment.
* Judgment by the investigator that the patient should not participate in the study if the patient is unlikely to comply with study procedures, restrictions, and requirements.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 100 (Estimated)
Dates: Start 2025-07-15 (Estimated); Primary Completion 2027-01-13 (Estimated); Study Completion 2027-01-13 (Estimated)

PRIMARY OUTCOMES:
Number of Participants with Grade 3 or greater Treatment Emergent Adverse Events (TEAEs) | Up to 25 weeks

SECONDARY OUTCOMES:
Number of Participants with any TEAEs | Up to 25 weeks
Number of Participants with Serious Adverse Events (SAEs), treatment related Adverse Events (AEs), treatment related SAEs, treatment related fatal AEs, non-fatal SAEs | Up to 25 weeks
Number of Participants with AEs leading to discontinuation of treatment, AEs leading to death, AEs leading to study withdrawal and AEs leading to dose modification | Up to 25 weeks
Change from baseline in hematology parameters: neutrophils, lymphocytes, monocytes, eosinophils, basophils and platelet count (Giga cells per Liter) | Baseline (Day 1) up to 25 weeks
Change from baseline in hematology parameter: Red Blood Cell (RBC) count (Trillion cells per Liter) | Baseline (Day 1) up to 25 weeks
Change from baseline in hematology parameter: Hemoglobin (Hb) (Grams per Liter) | Baseline (Day 1) up to 25 weeks
Change from baseline in hematology parameter: Reticulocytes (Percentage of reticulocytes) | Baseline (Day 1) up to 25 weeks
Change from baseline in hematology parameter: Mean Corpuscular Volume (MCV) (Femtoliters) | Baseline (Day 1) up to 25 weeks
Change from baseline in hematology parameter: Mean Corpuscular Hemoglobin (MCH) (Picograms) | Baseline (Day 1) up to 25 weeks
Change from baseline in clinical chemistry parameters: Blood urea nitrogen [BUN], glucose, calcium, sodium, and potassium levels (Millimoles per Liter) | Baseline (Day 1) up to 25 weeks
Change from baseline in clinical chemistry parameters: Total bilirubin, direct bilirubin and creatinine levels (Micromoles per Liter) | Baseline (Day 1) up to 25 weeks
Change from baseline in clinical chemistry parameters: Total protein levels (Gram per liter) | Baseline (Day 1) up to 25 weeks
Change from baseline in clinical chemistry parameters: Aspartate aminotransferase (AST), alanine aminotransferase (ALT) and alkaline phosphatase (ALP) levels (International units per liter) | Baseline (Day 1) up to 25 weeks
Change from Baseline in Vital signs: systolic blood pressure (SBP) and diastolic blood pressure (DBP) (Millimeters of mercury [mmHg]) | Baseline (Day 1) up to 25 weeks
Change from Baseline in Vital signs: pulse rate (Beats per minute) | Baseline (Day 1) up to 25 weeks
Change from Baseline in Vital signs: body temperature (Degrees Celsius) | Baseline (Day 1) up to 25 weeks
Change from Baseline in Vital signs: respiratory rate (breaths per minute) | Baseline (Day 1) up to 25 weeks
Change from Baseline in electrocardiogram (ECG) values: Heart rate (Beats per minute) | Baseline (Day 1) up to 25 weeks

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to anonymized individual patient-level data (IPD) and related study documents of the eligible studies via the Data Sharing Portal. Details on GSK's data sharing criteria can be found at: https://www.gsk.com/en-gb/innovation/trials/data-transparency/
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Anonymized IPD will be made available within 6 months of publication of primary, key secondary and safety results for studies in product with approved indication(s) or terminated asset(s) across all indications.
Access Criteria: Anonymized IPD is shared with researchers whose proposals are approved by an Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension may be granted, when justified, for up to 6 months.
URL: https://www.gsk.com/en-gb/innovation/trials/data-transparency/